CLINICAL TRIAL: NCT01047839
Title: Immunogenicity and Safety of the Japanese Encephalitis Vaccine IC51 (IXIARO®, JESPECT®) in a Pediatric Population in Non-endemic Countries. Uncontrolled, Open-label Phase 3 Study
Brief Title: Immunogenicity and Safety of the Japanese Encephalitis Vaccine IC51 (IXIARO®, JESPECT®) in a Pediatric Population in Non-endemic Countries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IC51-322
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Encephalitis
Keywords: Pediatric; Japanese Encephalitis Vaccine; non-endemic countries; to assess immunogenicity of purified inactivated Japanese Encephalitis (JE) vaccine IC51
MeSH Terms: conditions — Encephalitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- >=2 months to <3 years (Experimental): IC51 0.25 ml, 2 i.m. vaccinations at Day 0 and 28
  Interventions: Biological: IC51
- >=3 to <12 years (Experimental): IC51, 0.5 ml, 2 i.m. vaccinations at Day 0 and 28
  Interventions: Biological: IC51
- >=12 to <18 years (Experimental): IC51, 0.5 ml, 2 i.m. vaccinations at Day 0 and 28
  Interventions: Biological: IC51

INTERVENTIONS:
Biological: IC51 — 0.25 ml, 2 i.m. vaccinations at Day 0 and 28
  Arms: >=2 months to <3 years
Biological: IC51 — 0.5 ml, 2 i.m. vaccinations at Day 0 and 28
  Arms: >=12 to <18 years
Biological: IC51 — 0.5 ml, 2 i.m. vaccinations at Day 0 and 28
  Arms: >=3 to <12 years

SUMMARY:
The primary objective is to assess the safety profile of IC51 in a pediatric population from regions where JEV is not endemic

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy children and adolescents aged >=2 months to <18 years at the time of first vaccination
* Written informed consent by the subject's legal representative(s), according to local requirements, and written informed assent of the subject, if applicable
* Female subjects: either no childbearing potential or negative pregnancy test. For females after menarche willingness to practice a reliable method of contraception.
* The subject is planning to travel to an area where JE is endemic after completion of the vaccination schedule. Exposure to JE should be avoided until 1 week after the second IC51 dose and subjects should return from travel to JE endemic areas before the Month 7 visit. The planned travel to JE endemic areas should not interfere with the study visits and can take place between Visit 2 + 7 days to Month 7.

Exclusion Criteria:

* Clinical manifestation or history of any Flavivirus disease
* Vaccination against JE (except within this protocol), Yellow fever, West Nile virus and Dengue at any time prior or during the study
* History of immunodeficiency or immunosuppressive therapy
* Known HIV, HBV or HCV infection
* History of hypersensitivity reactions to other vaccines
* Acute febrile infection at each visit during which the subject receives a vaccination
* Active or passive immunization within 1 week before and 1 week after each IC51 vaccination.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ayad, Dr., Study Chair — Valneva Austria GmbH
Locations (10):
- United States (4):
  - Tampa Clinical Research Inc., Tampa, Florida
  - Passport Health, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Bronx Lebanon Hospital Center, New York, New York
- Australia (2):
  - Dr. Deb - The Travel Doctor, Brisbane, Queensland
  - Travel Doctor - TMVC Australia, Melbourne, Victoria
- Danske Laegers Forsknings Center, Søborg, Denmark
- Germany (2):
  - Berliner Zentrum für Reise- und Tropenmedizin, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- City Akuten Wasa Vaccination, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- >=2 Months to <3 Years: IC51 0.25 ml, 2 intramuscular vaccinations at Day 0 and Day 28
- >=12 to <18 Years: IC51, 0.5 ml, 2 intramuscular vaccinations at Day 0 and 28
Period: Overall Study
Arm/Group | >=2 Months to <3 Years | >=3 to <12 Years | >=12 to <18 Years
Started | 12 | 29 | 59
Completed | 10 | 29 | 53
Not Completed | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- >=2 Months to <3 Years: IC51 0.25 ml, 2 i.m.vaccinations at Day 0 and Day 28
- Total: Total of all reporting groups
Arm/Group | >=2 Months to <3 Years | >=3 to <12 Years | >=12 to <18 Years | Total
Number analyzed (Participants) | 12 | 29 | 59 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.81 (0.811) | 6.98 (2.417) | 15.90 (1.176) | 11.62 (5.605)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 36 | 53
  Male | 7 | 17 | 23 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 8 | 22 | 53 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Subjects With Serious Adverse Events (SAEs) and Medically Attended AEs up to Day 56 After the First Vaccination
Description: Rate of subjects with serious adverse events (SAEs) and medically attended AEs up to Day 56 after the first vaccination.
Time Frame: until Day 56
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- >=2 Months to <3 Years: IC51 0.25 ml, 2 i.m. vaccinations at Day 0 and Day 28
Arm/Group | >=2 Months to <3 Years | >=3 to <12 Years | >=12 to <18 Years
Number analyzed (Participants) | 12 | 29 | 59
percentage of participants | 33.3 [9.9 to 65.1] | 20.7 [8.0 to 39.7] | 3.4 [0.4 to 11.7]

2. Secondary Outcome: Rate of Subjects With Serious Adverse Events (SAEs) and Medically Attended AEs up to Month 7 After the First Vaccination
Time Frame: up to Month 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- IC51 0.25 mL: 0.25 mL i.m. vaccinations on Day 0 and Day 28 subjects aged >= 2 months to < 3years
- IC51 0.5 mL: 0.5 mL i.m. vaccinations on Day 0 and Day 28 subjects >= 3 years to < 18 years
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 12 | 88
percentage of participants
  SAEs | 0 [0.0 to 26.5] | 3.4 [0.7 to 9.6]
  medically attended AEs | 33.3 [9.9 to 65.1] | 18.2 [10.8 to 27.8]

3. Secondary Outcome: Rate of Subjects With Solicited Local and Systemic aEs Assessed With a Subject Diary for 7 Consecutive Days After Each Vaccination
Time Frame: 7 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 12 | 88
percentage of participants
  any Local after 1st Vaccination | 28.6 [2.1 to 48.4] | 48.9 [38.1 to 59.8]
  any Systemic after 1st Vaccination | 33.3 [2.1 to 48.4] | 46.0 [34.8 to 56.4]
  any Local after 2nd Vaccination | 22.2 [2.3 to 51.8] | 29.4 [20.0 to 40.3]
  any Systemic after 2nd Vaccination | 28.6 [2.3 to 51.8] | 22.6 [14.0 to 32.7]

4. Secondary Outcome: Rate of Subjects With Unsolicited AEs up to Day 56 and up to Month 7 After the First Vaccination
Time Frame: up to Day 56 and upt to Month 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 12 | 88
percentage of participants
  any unsolicited AE up to Day 56 | 83.3 [51.6 to 97.9] | 29.5 [20.3 to 40.2]
  any unsolicited AE up to Month 7 | 91.7 [61.5 to 99.8] | 43.2 [32.7 to 54.2]

5. Secondary Outcome: Rate of Subjects With Abnormal Laboratory Parameters up to Day 56 and up to Month 7 After the First Vaccination
Description: Laboratory parameters were assessed at the Day 28, Day 56 and Month 7 visit. Endpoint reflects abnormal laboratory parameters assessed as clinically significant by the investigator.
Time Frame: up to Month 7
Population: not from all subjects samples were collected, Overall number of participants analyzed were number of participants at Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 12 | 88
Participants
  White Blood cells on Day 28: number analyzed (Participants) | 8 | 83
  White Blood cells on Day 28 | 1 | 0
  Platelets on Day 28: number analyzed (Participants) | 8 | 83
  Platelets on Day 28 | 0 | 1

6. Secondary Outcome: SCRs as Defined as Percentage of Subjects With JEV Neutralizing Antibody Titers of PRNT 50 >= 1:10 at Day 56 and Month 7, Measured Using a Validated Plaque Reduction Neutralization Test (PRNT)
Time Frame: at Day 56 and Month 7
Population: number analyzed = number of subjects achieving seroconversion Overall number of participants analyzed were number of participants at Day 0
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 12 | 88
percentage of participants
  SCR Day 56: number analyzed (Participants) | 5 | 57
  SCR Day 56 | 100.0 [56.6 to 100.0] | 100.0 [93.7 to 100.0]
  SCR Month 7: number analyzed (Participants) | 2 | 32
  SCR Month 7 | 100.0 [34.2 to 100.0] | 90.6 [75.8 to 96.8]

7. Secondary Outcome: GMTs for JEV Neutralizing Antibodies Measured Using a Validated PRNT at Day 56 and Month 7
Time Frame: at Day 56 and Month 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | IC51 0.25 mL | IC51 0.5 mL
Number analyzed (Participants) | 5 | 59
Titer
  GMT Day 56 | 216.18 [105.97 to 441.00] | 340.74 [269.83 to 430.28]
  GMT Month 7 | 47.96 [0.00 to 3214485.72] | 57.12 [38.41 to 84.94]

8. Secondary Outcome: SCRs at Day 56 and Month 7 Stratified According to Dose Groups and Age Groups
Time Frame: at Day 56 and Month 7
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | >=2 Months to <3 Years | >=3 to <12 Years | >=12 to <18 Years
Number analyzed (Participants) | 12 | 29 | 59
percentage of participants
  SCR Day 56: number analyzed (Participants) | 5 | 15 | 42
  SCR Day 56 | 100 [56.6 to 100.0] | 100.0 [79.6 to 100.0] | 100.0 [91.6 to 100.0]
  SCR Month 7: number analyzed (Participants) | 2 | 3 | 29
  SCR Month 7 | 100.0 [34.2 to 100.0] | 66.7 [20.8 to 93.9] | 93.1 [78.0 to 98.1]

9. Secondary Outcome: GMTs at Day 56 and Month 7 Stratified According to Age Groups
Time Frame: at Day 56 and Month 7
Measure: Mean (95% Confidence Interval); unit: Titer
Arm/Group | >=2 Months to <3 Years | >=3 to <12 Years | >=12 to <18 Years
Number analyzed (Participants) | 5 | 15 | 42
Titer
  GMT Day 56 | 216.18 [105.97 to 441.0] | 508.03 [267.76 to 963.90] | 295.44 [235.96 to 369.90]
  GMT Month 7 | 47.96 [0.00 to 3214485.72] | 31.96 [0.48 to 2120.78] | 60.65 [40.72 to 90.36]

ADVERSE EVENTS:
Arm/Group | >=2 Months to <3 Years | >=3 to <12 Years | >=12 to <18 Years
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/29 | 3/59
Other Adverse Events (participants affected / at risk) | 11/12 | 22/29 | 49/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | >=2 Months to <3 Years (N=12) | >=3 to <12 Years (N=29) | >=12 to <18 Years (N=59)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | >=2 Months to <3 Years (N=12) | >=3 to <12 Years (N=29) | >=12 to <18 Years (N=59)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 2 (3) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 3 (5) | 2 (3) | 1 (1)
Influenza like Illness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 0 (0)
Ear Canal Erythema (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Initial Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Orapharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Injection Site Pain (General disorders) | 0 (0) | 3 (3) | 19 (25) — solicited local
Injection Site Itching (General disorders) | 0 (0) | 1 (1) | 3 (3) — solicited local
Tenderness (General disorders) | 1 (1) | 13 (19) | 31 (42) — solicited local
Hardening (General disorders) | 1 (2) | 0 (0) | 4 (4) — solicited local
Redness (General disorders) | 3 (3) | 2 (2) | 2 (2) — solicited local
Irritability (General disorders) | 0 (0) | 5 (7) | 1 (1) — solicited systemic
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (7) — solicited systemic
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) — solicited systemic
Excessive Fatigue (General disorders) | 0 (0) | 3 (3) | 7 (7) — solicited systemic
Muscle Pain (General disorders) | 0 (0) | 4 (5) | 23 (29) — solicited systemic
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1) — solicited systemic
Headache (Nervous system disorders) | 0 (0) | 3 (5) | 4 (8) — solicited systemic
Loss of appetite (General disorders) | 1 (1) | 1 (1) | 0 (0) — solicited systemic
Fever (General disorders) | 0 (0) | 1 (1) | 3 (3) — solicited systemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other